CLINICAL TRIAL: NCT07373327
Title: A Randomized Clinical Trial to Compare the Efficacy of Vinegar Dressing Versus Normal Saline Dressing in the Treatment of Diabetic Foot Ulcers
Brief Title: Vinegar vs Normal Saline Dressing for Diabetic Foot Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. MIAN MUHAMMAD BILAL, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp133
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer (DFU)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinegar Dressing (Experimental)
  Interventions: Other: Vinegar Dressing
- Normal Saline Dressing (Active Comparator)
  Interventions: Other: Normal Saline Dressing

INTERVENTIONS:
Other: Vinegar Dressing — In this arm, participants will receive a dressing made by soaking gauze in a vinegar solution. The solution will be prepared by adding one tablespoon of plain white vinegar to a cup of normal saline. The gauze will be applied to the wound in a wet-to-dry manner, twice daily, until the wound is fully healed or cultured negative. The goal is to assess the effectiveness of vinegar in promoting wound healing, reducing infection, and removing necrotic tissue.
  Arms: Vinegar Dressing
Other: Normal Saline Dressing — In this arm, participants will receive a dressing using normal saline (saltwater). The wound will be washed with normal saline and dressed in a wet-to-dry manner, twice daily, until the wound is fully healed or cultured negative. This arm will serve as the control group, with the goal of comparing the outcomes of saline dressing to vinegar dressing in terms of wound healing, bacterial infection reduction, and necrotic tissue removal.
  Arms: Normal Saline Dressing

SUMMARY:
This study is investigating the effectiveness of two different types of wound dressings in treating diabetic foot ulcers (DFUs), a common complication of diabetes that can be difficult to heal. The study will compare the use of vinegar dressings to normal saline (saltwater) dressings to see which one helps heal the wound faster and more effectively.

People with diabetic foot ulcers often struggle with infections and slow healing. The goal of this study is to determine if vinegar, a simple and affordable treatment, works better than saline in improving wound healing and reducing infections. The study will measure how quickly the wound heals, how much dead tissue is removed, and whether the bacteria in the wound disappear.

This study will involve patients with infected diabetic foot ulcers. Participants will be randomly assigned to receive either vinegar or saline dressing. The results will help determine the best and most cost-effective treatment for diabetic foot ulcers, potentially making it easier for patients to access better care.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 65 years.
* Gender: Both male and female participants are included.
* Condition: Patients with Grade 3 and 4 infected diabetic foot ulcers (DFU) according to the Wagner classification.

Exclusion Criteria:

* Wagner Grades 1, 2, 5, and 6 diabetic foot ulcers.
* History of Radiotherapy.
* History of Chemotherapy.
* Use of Steroids.
* Use of Immunosuppressive drugs.
* Allergy to vinegar.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Negative Cultures | From enrollment to 8 weeks after treatment initiation
  Definition: The proportion of participants whose wound cultures become negative (no bacterial growth) by the end of the treatment period (e.g., 3 weeks or 8 weeks).
  Measurement: The swab cultures will be taken weekly, and the presence or absence of bacterial infection will be recorded until the wound is culture-negative.
  Rationale: This outcome is crucial as it directly measures the effectiveness of vinegar dressing in reducing wound infection compared to normal saline dressing.

IPD SHARING:
Plan to Share IPD: Undecided